CLINICAL TRIAL: NCT07209475
Title: A Randomized Controlled Multicenter Trial, Examining the Effect of Amnio-Maxx on the Healing Rate of Chronic Diabetic Foot Ulcers.
Brief Title: Effect of Amnio-Maxx on the Healing Rate of Chronic Diabetic Foot Ulcers.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Royal Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Amnio-Maxx®
Record Dates: First submitted 2025-10-02; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Diabetic Foot Ulcer (DFU); Amnio-Maxx
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (Experimental): Cleansing, debridement, wound documentation, off-loading
  Interventions: Other: Standard of Care (Investigator Choice)
- Amnio-Maxx® Dual Layer Amnion Patch (Experimental): Application of Amnio-Maxx® Dual Layer Amnion Patch
  Interventions: Biological: Amnio-Maxx® Dual Layer Amnion Patch; Other: Standard of Care (Investigator Choice)

INTERVENTIONS:
Biological: Amnio-Maxx® Dual Layer Amnion Patch — Application of Amnio-Maxx® Dual Layer Amnion Patch
  Arms: Amnio-Maxx® Dual Layer Amnion Patch
Other: Standard of Care (Investigator Choice) — Cleansing, debridement, wound documentation, off-loading

SUMMARY:
This study will evaluate a cellular, acellular, matrix-like product (CAMP) and Standard of Care (SOC) versus SOC alone in the closure of nonhealing diabetic foot ulcers (DFUs). The study will evaluate Amnio-Maxx® Dual Layer Amnion Patch.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects are required to meet all the following criteria for enrollment into the study and subsequent randomization.

1. The potential subject is 18 years of age or older. At least 50% of the enrolled population must be > 65 years of age.
2. The potential subject has a history of Type I or Type II Diabetes Mellitus requiring treatment by a physician with either oral medications and/or insulin replacement therapy.
3. Potential subjects have an ulcer characterized by the following:

   1. Presence of a diabetic foot ulcer Wagner 1 or 2 grade at the first screening visit on any aspect of the foot, provided it is at or below the aspect of the medial malleolus. [NOTE: If two or more DFUs are present with the same grade, the index ulcer is the largest ulcer and the only one evaluated in the study. Index ulcer must be more than 5 cm distant apart.]
   2. A diabetic foot ulcer present for greater than 4 weeks (documented in the medical record) but less than 12 months duration if being treated with active SOC.
4. Objectively, less than 20% healing in the two-week screening period prior to randomization.
5. Study ulcer is a minimum of 1.0cm2 and a maximum of 25 cm2 post-debridement at first treatment visit.
6. Index ulcer and/or index ulcer limb may have had prior infection, but infection(s) must be adequately treated and controlled as defined by IDSA Guidelines Grade level 1
7. The subject is able and willing to follow the protocol requirements.
8. Subject has signed informed consent. Adequate circulation to the affected foot as demonstrated by a dorsum transcutaneous oxygen measurement (TCOM) or a skin perfusion pressure (SPP) measurement of ≥ 30 mmHg; an ABI between 0.7 and ≤ 1.3, or TBI of >6 within 3 months of the first Screening Visit.

10. Negative pregnancy test for females of childbearing potential (e.g., not post- menopausal for at least one year or surgically sterile). Females of childbearing potential must be willing to use acceptable methods of contraception (birth control methods, barriers, or abstinence) starting at Screening and continuing through the duration of their study participation.

11. The index ulcer has been offloaded with protocol defined offloading device throughout the study run-in period for at least 14 days prior to randomization (Run-in period defined as Screening through TV1/Randomization).

12. The index ulcer has a clean base and is free of necrotic debris at time of placement of treatment product.

Exclusion Criteria:

1. The Subject has a known life expectancy of < 1 year.
2. Index ulcer has been present for >1 year.
3. Patient does not have adequate 2-week historical data demonstrating < 20% area reduction.
4. Subject is unable to comply with offloading device.
5. Presence of any condition(s) which seriously compromises the subject's ability to complete this study or has a known history of poor adherence to medical treatment.
6. Subject has ulcers that are completely necrotic or fibrotic tissue
7. Subject has major uncontrolled medical disorders such as serious cardiovascular, renal, liver or pulmonary disease, lupus, palliative care or sickle cell anemia.
8. Subject currently being treated for an active malignant disease
9. or subjects with history of malignancy within the ulcer.
10. The Subject has other concurrent conditions that in the opinion of the Principal Investigator may compromise subject safety.
11. Known contraindications to amniotic tissue membranes or known allergies to any of the Amnio-Maxx components.
12. Concurrent participation in another clinical trial that involves an investigational drug or device that would interfere with this study.
13. Index ulcer has reduced in area by 20% or more after 2 weeks of standard of care from the first screening visit (S1) to the TV1/randomization visit.
14. Subject is pregnant or breastfeeding.
15. Subjects with a history of more than two weeks treatment with immunosuppressants (including systemic corticosteroids
16. >10mg daily dose), cytotoxic chemotherapy, or application of topical steroids to the ulcer surface within 30 days prior to randomization visit or who receive such medications during the screening period, or who are anticipated to require such medications during the course of the study.
17. Index ulcer has been previously treated with tissue engineered materials (e.g. Apligraf® or Dermagraft®) or other scaffold materials (e.g. Oasis, Matristem) within the last 30 days preceding the first treatment visit.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2026-08-14 (Estimated); Study Completion 2026-08-14 (Estimated)

PRIMARY OUTCOMES:
Complete Ulcer Closure | 12 weeks
Expected percentage area reduction (PAR) | 12-weeks

SECONDARY OUTCOMES:
Average percentage change from baseline in pain level related to the ulcer estimated from observed data using Numeric Pain Rating Scale (NPRS) and a Bayesian mixed effect model. | 12 weeks
Adverse events (AE) | 12 weeks

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Lion Heart Clinical Research, Burbank, California
  - Royal Research South, Miami, Florida
  - Denali Health Atlanta, LLC, Stone Mountain, Georgia
  - SerenaGroup Research Center, Omaha, Nebraska
  - Suffolk Foot and Ankle, East Patchogue, New York
  - Wound Care of Tulsa, Tulsa, Oklahoma
  - VAST Clinical Research Carrollton Foot Center, Carrollton, Texas
  - Elite Foot & Ankle Associates, Spicewood, Texas